CLINICAL TRIAL: NCT01091467
Title: Prospective Study of Heart Failure With Preserved Left Ventricular Ejection Fraction: Prevalence, Characterisation and Prognostic Significance of Cardiac Desynchrony
Brief Title: Prospective Study of Heart Failure With Preserved Left Ventricular Ejection Fraction
Acronym: KaRen
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Principal Investigator, Donal Erwan, Assistant Professor, French Cardiology Society
Other Study IDs: 08140
Record Dates: First submitted 2010-03-08; First posted 2010-03-24 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Congestive Heart Failure; Left Ventricular Ejection Fraction; Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure; Ejection Fraction; Echocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with HF: Each patient seen in hospital emergency or for congestive heart failure and with an ejection fraction above 45%

SUMMARY:
The purpose of this study is to examine electrical and echocardiographic characteristics and prognosis of consecutive patients admitted with acute heart failure and diagnosed to have heart failure with preserved ejection fraction (HFPEF).

DETAILED DESCRIPTION:
* Time 0: Patients will be screened at the time of presentation to the hospital at participating centres
* Usually patients will be hospitalised for an acute dyspnea in relation with a pulmonary congestion. This congestion does not necessarily justify a hospitalization and for part of the patients a consultation and a dedicated treatment would be good enough to cure the symptoms.
* Thus, patients seen in emergency for a congestion and diagnosed or known to have a preserved left ventricular ejection fraction (LV EF > 45%) will be proposed to participate to the study.
* Patients meeting inclusion criteria will be invited back to the clinic in stable condition, approximately 4-8 weeks after the initial hospitalization.
* Time 4-8 weeks after initial hospitalisation (NOT after discharge): Comprehensive history-taking and examinations.
* Any information necessary for the study will be collected by the principal investigator in each participating center in a dedicated, secure, e-CRF. The access to the e-CRF will be restrictive to the only principal investigator of each center. The lonely other persons able to take look to the e-CRF are the study monitors.
* Time 6, 12, and 18 months: Follow up by phone call or review of charts or other records such as death registries. This part of the study will be performed by the CRAs in the French Society of Cardiology

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to the hospital with congestive heart failure, defined as:

  1. Clinical signs of heart failure

     Major criteria
     * Paroxysmal nocturnal dyspnea
     * Orthopnea
     * Jugular venous distension
     * Pulmonary crackling rales
     * 3rd heart sound
     * Cardiothoracic ratio > 0.5 on X-ray
     * Pulmonary oedema on X-ray

     Minor Criteria
     * peripheral oedema
     * nocturnal cough
     * dyspnoea at exercise
     * hepatomegaly
     * pleural effusion
     * tachycardia (defined as ≥ 100 beats per minute)

     Heart failure if: presence of 2 major criteria or 1 major + 2 minor criteria
  2. LVEF ≥ 45% by echocardiography within 72h
  3. BNP > 100 ng/L or NT-proBNP > 300 ng/L

     Exclusion Criteria:
* Evidence of primary hypertrophic or restrictive cardiomyopathy or systemic illness known to be associated with infiltrative heart disease
* Known cause of right heart failure not related to left ventricular dysfunction
* Pericardial constriction
* Clinically significant pulmonary disease, as evidenced by requirement of home oxygen.
* End-stage renal disease requiring dialysis
* Bi-ventricular pacemaker (CRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the hospital with congestive heart failure
Sampling Method: Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Death rate | 18 months
  Analyse survival (all-cause death)

SECONDARY OUTCOMES:
Hospitalization for HF | 18 months
  Hospitalization for Heart Failure
Cardiovascular death | 18 months
  Cardiovascular death

CONTACTS AND LOCATIONS:
Locations (2):
- Pontchaillou Hospital, Rennes, France
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Donal E, Lund LH, Linde C, Edner M, Lafitte S, Persson H, Bauer F, Ohrvik J, Ennezat PV, Hage C, Lofman I, Juilliere Y, Logeart D, Derumeaux G, Gueret P, Daubert JC. Rationale and design of the Karolinska-Rennes (KaRen) prospective study of dyssynchrony in heart failure with preserved ejection fraction. Eur J Heart Fail. 2009 Feb;11(2):198-204. doi: 10.1093/eurjhf/hfn025. PMID 19168519
- [Result] Donal E, Lund L, Linde C, Daubert JC; KaRen investigators. Is cardiac resynchronization therapy an option in heart failure patients with preserved ejection fraction? Justification for the ongoing KaRen project. Arch Cardiovasc Dis. 2010 Jun-Jul;103(6-7):404-10. doi: 10.1016/j.acvd.2010.01.009. Epub 2010 Jun 23. PMID 20800804
- [Result] Donal E, Lund LH, Oger E, Hage C, Persson H, Reynaud A, Ennezat PV, Bauer F, Sportouch-Dukhan C, Drouet E, Daubert JC, Linde C; KaRen Investigators. Baseline characteristics of patients with heart failure and preserved ejection fraction included in the Karolinska Rennes (KaRen) study. Arch Cardiovasc Dis. 2014 Feb;107(2):112-21. doi: 10.1016/j.acvd.2013.11.002. Epub 2013 Dec 30. PMID 24388161
- [Result] Lund LH, Donal E, Oger E, Hage C, Persson H, Haugen-Lofman I, Ennezat PV, Sportouch-Dukhan C, Drouet E, Daubert JC, Linde C; KaRen Investigators. Association between cardiovascular vs. non-cardiovascular co-morbidities and outcomes in heart failure with preserved ejection fraction. Eur J Heart Fail. 2014 Sep;16(9):992-1001. doi: 10.1002/ejhf.137. Epub 2014 Jul 21. PMID 25046483
- [Result] Donal E, Lund LH, Oger E, Hage C, Persson H, Reynaud A, Ennezat PV, Bauer F, Drouet E, Linde C, Daubert C; KaRen investigators. New echocardiographic predictors of clinical outcome in patients presenting with heart failure and a preserved left ventricular ejection fraction: a subanalysis of the Ka (Karolinska) Ren (Rennes) Study. Eur J Heart Fail. 2015 Jul;17(7):680-8. doi: 10.1002/ejhf.291. Epub 2015 May 29. PMID 26033771
- [Result] Donal E, Lund LH, Oger E, Reynaud A, Schnell F, Persson H, Drouet E, Linde C, Daubert C; KaRen investigators. Value of exercise echocardiography in heart failure with preserved ejection fraction: a substudy from the KaRen study. Eur Heart J Cardiovasc Imaging. 2016 Jan;17(1):106-13. doi: 10.1093/ehjci/jev144. Epub 2015 Jun 16. PMID 26082167
- [Result] Hage C, Lund LH, Donal E, Daubert JC, Linde C, Mellbin L. Copeptin in patients with heart failure and preserved ejection fraction: a report from the prospective KaRen-study. Open Heart. 2015 Nov 3;2(1):e000260. doi: 10.1136/openhrt-2015-000260. eCollection 2015. PMID 26568833
- [Result] Savarese G, Donal E, Hage C, Oger E, Persson H, Daubert JC, Linde C, Lund LH; KaRen investigators. Changes in natriuretic peptides after acute hospital presentation for heart failure with preserved ejection fraction: A feasible surrogate trial endpoint? A report from the prospective Karen study. Int J Cardiol. 2017 Jan 1;226:65-70. doi: 10.1016/j.ijcard.2016.10.035. Epub 2016 Oct 17. PMID 27788392
- [Result] Bosseau C, Donal E, Lund LH, Oger E, Hage C, Mulak G, Daubert JC, Linde C; KaRen investigators. The prognostic significance of atrial fibrillation in heart failure with preserved ejection function: insights from KaRen, a prospective and multicenter study. Heart Vessels. 2017 Jun;32(6):735-749. doi: 10.1007/s00380-016-0933-8. Epub 2016 Dec 27. PMID 28028584
- [Result] Hage C, Michaelsson E, Linde C, Donal E, Daubert JC, Gan LM, Lund LH. Inflammatory Biomarkers Predict Heart Failure Severity and Prognosis in Patients With Heart Failure With Preserved Ejection Fraction: A Holistic Proteomic Approach. Circ Cardiovasc Genet. 2017 Feb;10(1):e001633. doi: 10.1161/CIRCGENETICS.116.001633. PMID 28100627
- [Result] Donal E, Lund LH, Oger E, Bosseau C, Reynaud A, Hage C, Drouet E, Daubert JC, Linde C; KaRen Investigators. Importance of combined left atrial size and estimated pulmonary pressure for clinical outcome in patients presenting with heart failure with preserved ejection fraction. Eur Heart J Cardiovasc Imaging. 2017 Jun 1;18(6):629-635. doi: 10.1093/ehjci/jex005. PMID 28329385
- [Result] Nagy AI, Hage C, Merkely B, Donal E, Daubert JC, Linde C, Lund LH, Manouras A. Left atrial rather than left ventricular impaired mechanics are associated with the pro-fibrotic ST2 marker and outcomes in heart failure with preserved ejection fraction. J Intern Med. 2018 Apr;283(4):380-391. doi: 10.1111/joim.12723. Epub 2018 Feb 12. PMID 29430747
- [Result] Savarese G, Donal E, Hage C, Oger E, Persson H, Daubert JC, Linde C, Lund LH; KaRen investigators. Corrigendum to "Changes in natriuretic peptides after acute hospital presentation for heart failure with preserved ejection fraction: A feasible surrogate trial endpoint? A report from the prospective Karen study" [Int. J. Cardiol. 226 (2017) 65-70]. Int J Cardiol. 2018 Jun 15;261:240. doi: 10.1016/j.ijcard.2018.03.075. Epub 2018 Mar 27. No abstract available. PMID 29602583
- [Result] Faxen UL, Hage C, Donal E, Daubert JC, Linde C, Lund LH. Patient reported outcome in HFpEF: Sex-specific differences in quality of life and association with outcome. Int J Cardiol. 2018 Sep 15;267:128-132. doi: 10.1016/j.ijcard.2018.04.102. PMID 29957252
- [Result] Persson H, Donal E, Lund LH, Matan D, Oger E, Hage C, Daubert JC, Linde C; KaRen Investigators. Importance of structural heart disease and diastolic dysfunction in heart failure with preserved ejection fraction assessed according to the ESC guidelines - A substudy in the Ka (Karolinska) Ren (Rennes) study. Int J Cardiol. 2019 Jan 1;274:202-207. doi: 10.1016/j.ijcard.2018.06.078. Epub 2018 Jun 20. PMID 30049496
- [Result] Lofstrom U, Hage C, Savarese G, Donal E, Daubert JC, Lund LH, Linde C. Prognostic impact of Framingham heart failure criteria in heart failure with preserved ejection fraction. ESC Heart Fail. 2019 Aug;6(4):830-839. doi: 10.1002/ehf2.12458. Epub 2019 Jun 17. PMID 31207140
- [Result] Najjar E, Faxen UL, Hage C, Donal E, Daubert JC, Linde C, Lund LH. ST2 in heart failure with preserved and reduced ejection fraction. Scand Cardiovasc J. 2019 Feb;53(1):21-27. doi: 10.1080/14017431.2019.1583363. Epub 2019 Mar 8. PMID 30776920
- [Derived] Donal E, Thebault C, Lund LH, Kervio G, Reynaud A, Simon T, Drouet E, Nonotte E, Linde C, Daubert JC. Heart failure with a preserved ejection fraction additive value of an exercise stress echocardiography. Eur Heart J Cardiovasc Imaging. 2012 Aug;13(8):656-65. doi: 10.1093/ehjci/jes010. Epub 2012 Jan 29. PMID 22291430